CLINICAL TRIAL: NCT00210600
Title: Assessment of Early and Standard Intervention With PROCRIT (Epoetin Alfa) 120,000 Units Once Every Three Weeks (Q3W) in Patients With Cancer Receiving Chemotherapy.
Brief Title: Early and Standard Intervention With 120,000 Units of PROCRIT (Epoetin Alfa) Every Three Weeks in Patients Receiving Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR003196
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Anemia
Keywords: Anemia; Hemoglobin level
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: PROCRIT (Epoetin alfa)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of PROCRIT (Epoetin alfa) when administered at 120,000 Units once every three weeks by comparing early dosing (Hb 11g/dL-12g/dL) vs. standard dosing (Hb< 11g/dL).

DETAILED DESCRIPTION:
This is a randomized, open-label, multi-center study. Eligible patients will be identified during the screening phase. After randomization, the Treatment Phase will start at the Day 1, Week 1 visit. The entire study period will be up to 22 weeks, with the screening phase lasting up to two weeks, treatment for a maximum of 16 weeks, and safety follow-up for four weeks. The primary objective of this study is to obtain efficacy and safety data regarding PROCRIT (Epoetin alfa) administered at 120,000 units subcutaneously (sc) once every three weeks (q3w) in 2 patient groups with cancer and anemia receiving chemotherapy:

1. Early Intervention Group: PROCRIT (Epoetin alfa) treatment started at patient hemoglobin (Hb) >= 11.0 g/dL to <= 12.0 g/dL and
2. Standard Intervention Group: PROCRIT (Epoetin alfa) treatment started once patient hemoglobin drops to < 11 g/dL or has a Hb <11.0 g/dL at study entry.

For safety monitoring, all patients will be followed for adverse events, hemoglobin (Hb), hematocrit (Hct), blood chemistries and blood pressure measurements throughout the study. All eligible patients with hemoglobin < 12.0 g/dL will be randomized to receive Epoetin alfa injections (120,000 Units ) under the skin every 3 weeks for a maximum of 16 treatment weeks. Doses may be adjusted depending on the patients hemoglobin levels.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed diagnosis of non-myeloid malignancy
* Baseline hemoglobin (Hb) value of >= 11.0 g/dL and <= 12.0 g/dL
* No blood transfusions in the 28 days prior to the start of Treatment Phase
* Must be receiving chemotherapy or will begin receiving chemotherapy at start of Treatment
* Iron transferrin saturation (TSAT) > 20% or if TSAT<20%, serum ferritin must be greater than 100 ng/mL.

Exclusion Criteria:

* No myeloid malignancy or known history of myelodysplasia
* No planned radiation during the study
* Prior treatment with Epoetin alfa or any other erythropoietic agent (e.g., Darbepoetin alfa, gene-activated erythropoietin) within the previous three months
* No uncontrolled disease/dysfunction of the lung, cardiovascular, endocrine, neurologic, gastrointestinal, or genitourinary systems
* No history of uncontrolled cardiac arrhythmias (within 6 months) or pulmonary emboli, deep vein thrombosis, ischemic stroke, other arterial or venous thrombotic events (excluding superficial thromboses), or known history of chronic hypercoagulable disorders
* Has not received an experimental drug or device within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2005-05; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The proportion of weekly hemoglobin levels for all patients in each group during the 16 week PROCRIT (Epoetin alfa) treatment that are > 11.0 g/dL and < 13.0 g/dL.

SECONDARY OUTCOMES:
The proportion of patients in the early intervention group for whom all hemoglobin values during the 16 week PROCRIT (Epoetin alfa) treatment were > 11.0 g/dL and < 13.0 g/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Assessment of Early and Standard Intervention with PROCRIT (Epoetin alfa) 120,000 Units Once Every Three Weeks (Q3W) in Patients with Cancer Receiving Chemotherapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=506&filename=CR003196_CSR.pdf